CLINICAL TRIAL: NCT03188172
Title: MUK Nine b: OPTIMUM. A Phase II Study Evaluating Optimised Combination of Biological Therapy in Newly Diagnosed High Risk Multiple Myeloma and Plasma Cell Leukaemia.
Brief Title: MUK Nine b: OPTIMUM Treatment Protocol
Acronym: MUKnineb
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Myeloma UK (Other); Celgene (Industry); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM16/235
Record Dates: First submitted 2017-05-02; First posted 2017-06-15 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Bortezomib; Lenalidomide; daratumumab; Dexamethasone; Melphalan; Filgrastim

STUDY DESIGN:
Intervention Model Description: The trial is designed as a single arm phase II trial with interim assessments for futility, using a Bayesian strategy for monitoring multiple outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial Treatment (Experimental): Induction:
  Cyclophosphamide 500mg, days 1, 8 Bortezomib 1.3mg/m2, days 1, 4, 8, 11 Lenalidomide 25mg, days 1-14 Daratumumab 16mg/kg, days 1, 8, 15 (cycles 1& 2), day 1 only from cycle 3 Dexamethasone 20-40mg, days 1, 4, 8, 11
  ASCT stem cell harvest:
  with Bortezomib 1.3mg/m2, (12 hours post melphalan) Bortezomib 1.3mg/m2, day +5, +14, weekly
  Consolidation part 1:
  Bortezomib 1.3mg/m2 days 1, 8, 15, 22 Lenalidomide 25mg days 1-21 Daratumumab 16mg/kg day 1 Dexamethasone 20-40mg days 1, 8, 15, 22
  Consolidation part 2:
  Bortezomib 1.3mg/m2 days 1, 8, 15 Lenalidomide 25mg days 1-21 Daratumumab 16mg/kg day 1
  Maintenance:
  Lenalidomide 10mg days 1-21 Daratumumab 16mg/kg day 1
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Lenalidomide; Drug: Daratumumab; Drug: Dexamethasone; Drug: Melphalan; Drug: Filgrastim

INTERVENTIONS:
Drug: Cyclophosphamide — Chemotherapy
Drug: Bortezomib — Chemotherapy
  Other Names: Velcade
Drug: Lenalidomide — Chemotherapy
  Other Names: Revlamid
Drug: Daratumumab — Chemotherapy
  Other Names: Daralex
Drug: Dexamethasone — Chemotherapy
Drug: Melphalan — Chemotherapy
Drug: Filgrastim — Haematopoietic agent for the stem cell harvest

SUMMARY:
To determine whether a combination of four novel agents bortezomib(Velcade), lenalidomide (Revlimid), Daratumumab (Darzalex) & dexamethasone in combination with low-dose cyclophosphamide is sufficiently active in a high risk population of myeloma patients, to take forward into a phase III trial compared to standard treatment.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a plasma cell tumour with an annual incidence in the UK of approximately 40 -50 per million i.e. 4500 new cases per annum. Approximately 20% of the patients diagnosed with multiple myeloma have a significantly worse prognosis at 3 years than other multiple myeloma patients and these are characterised as having high risk (HR) disease defined by genetic lesions and gene expression profiles (GEP). There have been no significant improvements in outcome over the last decade for patients with HR disease. Therefore, it is important to identify more effective treatment options for this group of patients especially given that the number of novel agents are potentially available and which can be given as part of intensive therapy regimen.

Intensive treatment in HR patients has been used outside the UK with promising results but access to drugs in the UK has been challenging with constraints in the NHS treatment pathway. This is the first time in the UK that newly diagnosed multiple myeloma patients may be entered into a clinical trial prospectively according to their genetic risk profile. It provides a unique opportunity to improve outcomes and provide evidence for high cost novel treatment strategies in this restricted population of poor prognosis patients.

The MUKnine trial is designed to evaluate the novel treatment strategies for multiple myeloma patients with HR disease and incorporate a genetic screening component. Patients identified as having HR disease are then invited to take part in the phase II single arm, multi centre trial that investigates the intensive treatment schedule comprising four novel agents bortezomib (Velcade), lenalidomide (Revlimid), daratumumab (Daralex), dexamethasone with cyclophosphamide. The trial will determine if this treatment strategy is sufficiently active to take forward in to further testing in this population. Patients identified as not having HR disease will receive standard local treatment and will be followed up in a cohort study to assess response, progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of High Risk status from Institute of Cancer Research (ICR) following bone marrow and blood sample processed through the MUKnine a screening protocol.
2. Previously untreated participants, although participants may have received up to 2 cycles of cyclophosphamide, thalidomide, dexamethasone (CTD), cyclophosphamide, velcade, dexamethasone (CVD), cyclophosphamide, lenalidomide, dexamethasone (CRD) or velcade, thalidomide, dexamethasone (VTD) pre-trial induction chemotherapy while awaiting the results of the laboratory analysis from the MUKnine a Screening Protocol. (In addition, non-systemic therapy such as therapeutic plasma exchange, dexamethasone up to a maximum of 160mg or radiotherapy sufficient to alleviate or control pain or local invasion is permitted).
3. Measurable disease with at least one of the following or willing to undergo further bone marrows for assessment:

   - Paraprotein ≥ 5g/L or ≥ 0.5 g/L for IgD subtypes.

   - Serum free kappa or lambda light chains ≥ 100 mg/L with abnormal ratio (for light chain only myeloma).

   - Urinary Bence Jones protein ≥ 200 mg/L.
4. Non measurable participants providing they accept a 3 monthly bone marrow during induction and a 6 monthly bone marrow assessment during consolidation and maintenance.
5. Aged 18 years or over.
6. Fit for intensive chemotherapy and autologous stem cell transplant (at clinician's discretion).
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
8. The Celgene Pregnancy Prevention Plan must be followed and participants must agree to comply with this:

   * Females of childbearing potential (FCBP) must agree to utilise two reliable forms of contraception simultaneously or practice complete abstinence for at least for 28 days prior to starting trial treatment, during the trial and for at least 28 days after trial treatment discontinuation, and even in case of dose interruption, and must agree to regular pregnancy testing during this timeframe.
   * Males must agree to use a latex condom during any sexual contact with FCBP during the trial, including during dose interruptions and for 28 days following discontinuation from this trial even if he has undergone a successful vasectomy o Males must also agree to refrain from donating semen or sperm while on trial treatment including during any dose interruptions and for at least 6 months after discontinuation from this trial
   * All participants must agree to refrain from donating blood while on trial drug including during dose interruptions and for 28 days after discontinuation from this trial.
9. Calculated creatinine clearance ≥ 30mL/min (using Cockcroft-Gault formula).
10. Alanine transaminase (ALT) and/or Aspartate transaminase (AST) ≤ 2.5 times upper limit of normal (ULN).
11. Bilirubin ≤ 2.0 x ULN, except in participants with congenital bilirubinemia, such as Gilbert syndrome (direct bilirubin ≤2.0 times ULN
12. Platelet count ≥ 75 x 109/L. (≥ 50 x 109/L if myeloma involvement in the bone marrow is >50%). Platelet support is permitted.
13. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L. Growth factor support is permitted.
14. Haemoglobin ≥ 80 g/L. (Participants may be receiving red blood cell (RBC) transfusions in accordance with institutional guidelines.
15. Corrected serum calcium ≤ 3.5 mmol/L.

Exclusion Criteria:

1. Solitary bone/solitary extramedullary plasmacytoma.
2. Primary diagnosis of amyloidosis, monoclonal gammopathy of undetermined significance or smoldering multiple myeloma or Waldenstrom's Disease.
3. Prior or concurrent invasive malignancies except the following:

   * Adequately treated basal cell or squamous cell skin cancer.
   * Incidental finding of low grade (Gleason 3+3 or less) prostate cancer.
   * Any cancer from which the subject has been disease free for at least 3 years.
4. Known/underlying medical conditions that, in the investigator's opinion, would make the administration of the study drug hazardous (e.g. uncontrolled diabetes or uncontrolled coronary artery disease).
5. Any clinically significant cardiac disease, including:

   - myocardial infarction within 1 year before randomization, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV.

   - Uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4 Grade ≥2) or clinically significant ECG abnormalities.

   - screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec. · Known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume [FEV] in 1 second <60% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (intermittent asthma is allowed). Participants with known or suspected COPD or asthma must have a FEV1 test during screening.
6. Known to be seropositive for history of human immunodeficiency virus (HIV) or known to have active hepatitis B or hepatitis C.
7. Any known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts), or known sensitivity to mammalian-derived products.
8. Clinically significant allergies or intolerance to cyclophosphamide, lenalidomide, velcade, daratumumab or dexamethasone. · Previous treatment with daratumumab or any other anti-CD38 therapies.
9. Participants with contraindication to thromboprophylaxis.
10. Grade 2 or greater peripheral neuropathy (per NCI-CTCAEv4.0).
11. Participants with POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
12. Any concurrent medical or psychiatric condition or disease (e.g., active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
13. Known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder). Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
14. Participant is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this trial or within at least 6 months after the last dose of trial treatment. Or, participant is a man who plans to father a child while taking part in this trial or within at least 6 months after the last dose of trial treatment.
15. Major surgery within 2 weeks before treatment protocol registration or has not fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study. Kyphoplasty or vertebroplasty is not considered major surgery.
16. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before treatment protocol registration or is currently enrolled in an interventional investigational study.

Inclusion Criteria for ASCT

1. Minimum stem cell harvest of 2 x 106 CD34+ cells/kg body weight.
2. Received a minimum of 4, unless a complete response (CR) has been achieved with a lesser number, or a maximum of 6 Induction (CVRDd) cycles.
3. Achieved a response of stable disease (SD) or better.

Exclusion Criteria for ASCT 1. Participants that have progressive disease.

Inclusion Criteria for Consolidation Part 1 (VRDd)

1. Undergone autologous transplant with high dose melphalan-velcade (HDM-V) conditioning (Participants must have received a minimum of 100 mg/m2 Melphalan in order to proceed with consolidation).
2. Neutrophils ≥ 1.0 x 109/L. Growth factor support is permitted.
3. Platelet count ≥ 75 x 109/L. Platelet support is permitted.

Exclusion Criteria for Consolidation Part 1 (VRDd)

1. Participants that have progressive disease.

Inclusion Criteria for Consolidation Part 2 (VRD)

1. Received 6 cycles of Consolidation Part 1 (VRDd) or 1 cycle of VRd pre-harvest plus 5 cycles of Consolidation Part 1 (VRDd).
2. Neutrophils ≥ 1.0 x 109/L. Growth factor support is permitted.
3. Platelet count ≥ 75 x 109/L. Platelet support is permitted.

Exclusion Criteria for Consolidation Part 2 (VRD)

1. Participants that have progressive disease.

Inclusion Criteria for Maintenance (RD)

1. Received 12 cycles of Consolidation Part 2 (VRD).
2. Neutrophils ≥ 1.0 x 109/L. Growth factor support is permitted.
3. Platelet count ≥ 75 x 109/L. Platelet support is permitted.

Exclusion Criteria for Maintenance (RD)

1. Participants that have progressive disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | At 18 months post registration
  Defined as the time from registration until first documented evidence of progressive disease or death. Participants not progressed at analysis will be censored at the last date known to be alive and progression free.

SECONDARY OUTCOMES:
Occurrence of Serious Adverse Events(SAE) and Suspected, Unexpected Serious Adverse Reactions (SUSAR) | At 120 days post autologous stem cell transplant (ASCT)
  Will be reported based on occurrence of SAE & SUSARs with details of causality and expectedness.
Progression free survival at 100 days post autologous stem cell transplant | At 100 days post ASCT
  Determine whether the treatment schedule should be dropped for futility
Minimal residual disease (MRD) negative disease | At 100 days post ASCT
  Defined as absence of aberrant phenotype plasma cells
Overall survival | At 12 months, 24 months & 36 months post registration
  Median overall survival estimates
Maximum response | From registration to end of induction therapy, 100 days post ASCT, post consolidation part 2
  Proportion of participants achieving each response category. Time from registration until the participant achieves a maximum response.
Overall response | At end of induction therapy, 100 days post ASCT, post consolidation part 2
  Proportion of participants receiving at least a partial response
Second progression free survival | From registration until second disease progression, 3 years
  Time from registration to second disease progression or death.
Overall treatment benefit | At the end of induction therapy and 100 days post autologous stem cell transplant
  Clinician assessment of treatment benefit will be obtained
Quality of life using the EQ-5D questionnaire | From registration until second disease progression, 3 years
  Quality of life will be summarised at each post-registration timepoint, adjusting for baseline mean scores and 95% confidence intervals. This will also be summarised descriptively using bar charts, box plots, plots of mean QoL over time and summary tables.
Quality of life using the EORTC QLQ-C30 questionnaire | From registration until second disease progression, 3 years
  Quality of life will be summarised at each post-registration timepoint, adjusting for baseline mean scores and 95% confidence intervals. This will also be summarised descriptively using bar charts, box plots, plots of mean QoL over time and summary tables.
Quality of life using the QLQ-MY20 questionnaire | From registration until second disease progression, 3 years
  Quality of life will be summarised at each post-registration timepoint, adjusting for baseline mean scores and 95% confidence intervals. This will also be summarised descriptively using bar charts, box plots, plots of mean QoL over time and summary tables.

OTHER OUTCOMES:
Progression free survival (comparison with Myeloma XI/XI+ data) | From registration until second disease progression, 3 years
  Matched comparison of progression free survival
Impact of minimal residual disease on progression free survival | From registration until second disease progression, 3 years
  Analysis will include any participant with a MRD assessment
Genomic instability | From registration until second disease progression, 3 years
  To be investigated in an exploratory manner and will include analysis of new genetic abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaiser, Principal Investigator — University of Leeds
Locations (21):
- United Kingdom (21):
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Royal Hampshire County Hospital, Bournemouth
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology & Oncology Centre, Bristol
  - Ninewells Hospital, Dundee
  - Beatson Oncology Centre, Glasgow
  - Kettering General Hosptial, Kettering
  - Leicester Royal Infirmary, Leicester
  - Kings College Hosptial, London
  - Manchester Royal Infirmary, Manchester
  - The Christie Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hosptial, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Royal Stoke Hospital, Stoke-on-Trent
  - Royal Marsden Hospital, Sutton
  - Worcester Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keaveney S, Dragan A, Rata M, Blackledge M, Scurr E, Winfield JM, Shur J, Koh DM, Porta N, Candito A, King A, Rennie W, Gaba S, Suresh P, Malcolm P, Davis A, Nilak A, Shah A, Gandhi S, Albrizio M, Drury A, Pratt G, Cook G, Roberts S, Jenner M, Brown S, Kaiser M, Messiou C. Image quality in whole-body MRI using the MY-RADS protocol in a prospective multi-centre multiple myeloma study. Insights Imaging. 2023 Oct 15;14(1):170. doi: 10.1186/s13244-023-01498-3. PMID 37840055
- [Derived] Kaiser MF, Hall A, Walker K, Sherborne A, De Tute RM, Newnham N, Roberts S, Ingleson E, Bowles K, Garg M, Lokare A, Messiou C, Houlston RS, Jackson G, Cook G, Pratt G, Owen RG, Drayson MT, Brown SR, Jenner MW. Daratumumab, Cyclophosphamide, Bortezomib, Lenalidomide, and Dexamethasone as Induction and Extended Consolidation Improves Outcome in Ultra-High-Risk Multiple Myeloma. J Clin Oncol. 2023 Aug 10;41(23):3945-3955. doi: 10.1200/JCO.22.02567. Epub 2023 Jun 14. PMID 37315268
- [Derived] Rata M, Blackledge M, Scurr E, Winfield J, Koh DM, Dragan A, Candito A, King A, Rennie W, Gaba S, Suresh P, Malcolm P, Davis A, Nilak A, Shah A, Gandhi S, Albrizio M, Drury A, Roberts S, Jenner M, Brown S, Kaiser M, Messiou C. Implementation of Whole-Body MRI (MY-RADS) within the OPTIMUM/MUKnine multi-centre clinical trial for patients with myeloma. Insights Imaging. 2022 Jul 28;13(1):123. doi: 10.1186/s13244-022-01253-0. PMID 35900614
- [Derived] Oliva S, Kaiser MF. Is it time to tailor treatment on the basis of minimal residual disease in multiple myeloma? Lancet Haematol. 2021 Dec;8(12):e876-e877. doi: 10.1016/S2352-3026(21)00341-0. No abstract available. PMID 34826409
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481